CLINICAL TRIAL: NCT06925841
Title: The Effect of Mother-Baby Themed Coloring on Stress, Anxiety, and Psychosocial Health in Pregnant Women Diagnosed With Preeclampsia: A Randomized Controlled Trial
Brief Title: Psychosocial Effects of Coloring in Preeclamptic Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Collaborators: necmettin erbakan university Scientific Research Projects (BAP) (Unknown)
Responsible Party: Principal Investigator, Sibel Kıyak, Assist. Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023/425:14022
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Preeclampsia; Anxiety; Pregnancy; Stress
Keywords: preeclampsia; anxiety; pregnancy; mandala; stress; cortisol
MeSH Terms: conditions — Pre-Eclampsia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two groups with intervention group and control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mother and Baby Themed Coloring Activity (Experimental): Participants in this intervention group will color mother-and-baby-themed images provided by the researcher using a free coloring technique. In addition to routine care, each pregnant woman will participate in a structured 30-minute coloring activity each day.
  Interventions: Other: Experimental
- Routine care (Active Comparator): The patients in the control group will receive only routine care and treatment.
  Interventions: Other: routine care

INTERVENTIONS:
Other: Experimental — Two pre-selected mother-baby themed images to be used in the study will be printed separately on A4-sized papers (21.0 cm × 29.7 cm). Each participant will receive a new image every day.At the beginning of the study, each participant will be provided with a set of 12 colored pencils (orange, red, pink, purple, light blue, dark blue, light green, dark green, light brown, dark brown, black, and white). Colored pencils have been preferred over soft-tipped pencils due to their requirement for greater physical effort and their ability to facilitate a clearer expression of emotions. Participants in the intervention group will receive routine care and will engage in a 30-minute daily coloring activity.
  Arms: Mother and Baby Themed Coloring Activity
Other: routine care — The control group will receive routine care provided by the nurse.
  Arms: Routine care

SUMMARY:
Preeclampsia is one of the major causes of maternal and neonatal mortality and morbidity, affecting approximately 3-5% of pregnancies. A diagnosis of preeclampsia may lead to psychological problems such as psychosocial distress, depression, and anxiety due to prolonged hospitalization, concerns about the future health of the baby, separation from family, and adapting to a foreign environment. Health professionals play a crucial role in the diagnosis, treatment, and care of high-risk pregnancies and also implement non-pharmacological supportive methods such as yoga, progressive muscle relaxation, and mindfulness. One of these non-pharmacological methods is mandala. According to the literature, integrating mandala coloring into perinatal care is believed to have beneficial effects.

Therefore, the primary aim of this study is to investigate the effects of mother-baby themed coloring on anxiety. The secondary aim is to determine its effects on psychosocial health and cortisol levels.

H1a: Is there a difference between anxiety scores in preeclamptic pregnant women who were and were not exposed to dyeing activity?

H1b: Is there a difference between psychosocial health scores in preeclamptic pregnant women who were and were not exposed to dyeing activity?

H1c: Is there a difference between cortisol levels in preeclamptic pregnant women who were and were not exposed to dyeing activity?

ELIGIBILITY:
Inclusion Criteria:

* Having a single and healthy fetus
* Gestational age ≥ 20 weeks
* Diagnosed with preeclampsia by a physician
* Not having a history of treated pregnancy

Exclusion Criteria:

* Using psychiatric medication (self-report)
* Receiving psychological counseling during the intervention
* Diagnosed with severe preeclampsia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Anxiety | nine months
  The State-Trait Anxiety Inventory was used to determine the anxiety level. The scale consists of a total of 40 items, with 20 items for state anxiety and 20 items for trait anxiety. In this study, the state anxiety section of the scale will be used. The scale is a four-point Likert-type, with items scored between 1 and 4 (1 = not at all, 2 = a little, 3 = quite a bit, 4 = completely). The score range for each subscale is between 20 and 80 points. Items 1, 2, 5, 8, 10, 11, 15, 16, 19, 20, 21, 26, 27, 30, 33, 36, and 39 are positively worded and do not express anxiety. Therefore, these items are reverse coded during the analysis phase. As the score obtained from the scale increases, the level of anxiety also increases.

SECONDARY OUTCOMES:
Psychosocial health | nine months
  The Pregnancy Psychosocial Health Assessment Scale was used to evaluate psychosocial health during pregnancy. It consists of 46 items and has six subscales (characteristics related to pregnancy and partner relationship, characteristics related to anxiety and stress, characteristics related to domestic violence, characteristics related to psychosocial support needs, family characteristics, and characteristics related to physical-psychosocial changes in pregnancy). The total score obtained from the scale is divided by the number of items to determine the average value, resulting in a score between 1 and 5. The closer the total score is to 1, the greater the problem in psychosocial health during pregnancy, and a score of 1 indicates very poor psychosocial health. The same evaluation applies to the subscales, and the closer the score is to 1, the more likely there is a problem with that specific factor.
Cortisol | nine months
  Cortisol measurement will be conducted on Day 1 (pre-test) and Day 3 (post-test). To determine cortisol levels, blood samples will be collected from participants in both the intervention and control groups between 08:00 and 10:00 in the morning. Blood samples will be taken by nurses working in the clinic. Typically, the blood volume collected from each participant is 3-4 ml. The collected blood samples will be analyzed in the Biochemistry Laboratory of the Faculty of Medicine using the Electrochemiluminescence Immunoassay (ECLIA) method. Blood samples from both the intervention and control groups will be centrifuged at 4000 rpm for 10 minutes. Serum cortisol samples will be measured using the Cobas cortisol kit (Roche Diagnostics, USA) with the fully automated Roche Elecsys 8000 (Hitachi; Roche Diagnostics, Germany) device according to the ECLIA method.

CONTACTS AND LOCATIONS:
Overall Officials: Kamile Altuntuğ, Professor, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No